CLINICAL TRIAL: NCT07315282
Title: The Effect of Oral Iron Supplements on Insulin and Glucose Metabolism in Overweight and Obese Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicole Stoffel (Other)
Collaborators: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor-Investigator, Nicole Stoffel, Prof. Dr., ETH Zurich
Organization: ETH Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FIND
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Overweight and Obese Women
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-dose iron supplementation (Experimental): 195 mg iron as ferrous sulfate daily for 14 days
  Interventions: Dietary Supplement: 195 mg iron daily
- low-dose iron supplementation (Active Comparator): 15 mg iron as ferrous fumarate daily for 14 days
  Interventions: Dietary Supplement: 15 mg iron daily

INTERVENTIONS:
Dietary Supplement: 195 mg iron daily — 3 x 65 mg iron as ferrous sulfate
  Arms: high-dose iron supplementation
Dietary Supplement: 15 mg iron daily — 3 x 5 mg iron as ferrous sulfate
  Arms: low-dose iron supplementation

SUMMARY:
The study will be a randomized, double-blind, 17-day metabolic intervention trial including 14 days of high-dose or low-dose iron supplementation. A total of 70 overweight or obese (OW/OB) women will be enrolled. Participants will be individually randomized into either the high-iron or low-iron group.

Women in the low-iron group will receive 15 mg of iron as ferrous fumarate daily for 14 days, while women in the high-iron group will receive 195 mg of iron as ferrous sulfate daily for 14 days.

The study consists of three visits in total. On Day 0, a fasting blood sample will be collected and an OGTT will be performed, with additional blood samples collected at 1 hour and 2 hours post-OGTT. The OGTT will be repeated on Day 14, after 14 days of oral iron supplementation, and again on Day 17, four days after oral iron supplementation has been stopped

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 27.5 kg/m2
* serum ferritin <30 μg/L
* hemoglobin ≥ 11 g/dl
* fasting blood glucose < 5.6 mmol/L

Exclusion Criteria:

* intravenous or high dose oral iron in the preceding 2 months
* medical disorders are known to affect iron absorption or metabolism, or T2DM
* cigarette smoking
* recent blood transfusion or major blood loss

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-23 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood glucose increase during OGTT Day 0 | Day 0
  Blood glucose increase during OGTT before the intake of oral iron for 14 days
Blood glucose increase during OGTT Day 14 | Day 14
  Blood glucose increase during OGTT after the intake of oral iron for 14 days

SECONDARY OUTCOMES:
Insulin increase during OGTT Day 0 | Day 0
  Insulin increase during OGTT before the intake of oral iron for 14 days
Insulin increase during OGTT Day 14 | Day 14
  Insulin increase during OGTT after the intake of oral iron for 14 days
Serum Hepcidin Day 0 | Day 0
  Serum Hepcidin measured before the intake of oral iron
Serum Hepcidin D14 | Day 14
  Serum Hepcidin measured after the intake of oral iron
Serum Ferritin Day 0 | Day 0
  Serum Ferritin measured before the intake of oral iron
Serum Ferritin Day 14 | Day 14
  Serum Ferritin measured after the intake of oral iron
Soluble Transferrin Receptor (sTfR) Day 0 | Day 0
  sTfR measured before the intake of oral iron
Soluble Transferrin Receptor (sTfR) Day 14 | Day 14
  sTfR measured after the intake of oral iron
Hemoglobin Day 0 | Day 0
  Hemoglobin measured before the intake of oral iron
Hemoglobin Day 14 | Day 14
  Hemoglobin measured after the intake of oral iron
C-reactive protein (CRP) Day 0 | Day 0
  CRP measured before the intake of oral iron
C-reactive protein (CRP) Day 14 | Day 14
  CRP measured after the intake of oral iron
Alpha-1-acid glycoprotein (AGP) Day 0 | Day 0
  AGP measured before the intake of oral iron
Alpha-1-acid glycoprotein (AGP) Day 14 | Day 14
  AGP measured after the intake of oral iron
Serum Iron Day 0 | Day 0
  Serum Iron measured before the intake of oral iron
Serum Iron Day 14 | Day 14
  Serum Iron measured after the intake of oral iron
Total Iron Binding Capacity (TIBC) Day 0 | Day 0
  TIBC measured before the intake of oral iron
Total Iron Binding Capacity (TIBC) Day 14 | Day 14
  TIBC measured after the intake of oral iron
Transferrin Saturation (TSAT) Day 0 | Day 0
  TSAT measured before the intake of oral iron
Transferrin Saturation (TSAT) Day 14 | Day 14
  TSAT measured after the intake of oral iron
Transferrin Saturation (TSAT) Day 17 | Day 17
  TSAT measured at endpoint
Total Iron Binding Capacity (TIBC) Day 17 | Day 17
  TIBC measured at endpoint
Serum Iron Day 17 | Day 17
  Serum Iron measured at endpoint
Serum Hepcidin Day 17 | Day 17
  Serum Hepcidin measured at endpoint
Insulin increase during OGTT Day 17 | Day 17
  Insulin increase during OGTT at Endpoint
Blood glucose increase during OGTT Day 17 | Day 17
  Blood glucose increase during OGTT at Endpoint
Fasting blood glucose Day 0 | Day 0
  Fasting blood glucose before iron intake
Fasting blood glucose Day 14 | Day 14
  Fasting blood glucose after iron intake
Fasting blood glucose Day 17 | Day 17
  Fasting blood glucose at Endpoint
Fasting insulin Day 0 | Day 0
  Fasting insulin before iron intake
Fasting insulin Day 14 | Day 14
  Fasting insulin after iron intake
Fasting insulin Day 17 | Day 17
  Fasting insulin at Endpoint
Blood glucose profile measured over the 14 days | Day 0 - Day 14
  blood glucose profile measured by wearable FreeStyle Libre Sensor

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No